CLINICAL TRIAL: NCT04733937
Title: Protocol Title: Comparative Effects of A2 Platinum® Stage 1 Infant Formula Versus Conventional Stage 1 Infant Formula Containing A1 and A2 Β-casein Versus Breast Feeding on Infant Digestion and Comfort: a Single-blind Randomized Controlled Trial
Brief Title: Comparative Effects of A2 Platinum Stage 1 Infant Formula on Infant Digestion and Comfort
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: a2 Milk Company Ltd. (Industry)
Collaborators: Shanghai First Maternity and Infant Hospital (Other); Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Edanz Group Japan Ltd (Unknown); Women & Children's Health Care Hospital of Linyi, China (Unknown); Beijing Esmile Technology Co. Ltd. (Unknown); Nanjing Maternity and Child Health Care Hospital (Other); First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other); Second Hospital of Jilin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: A2MC-G190549140
Record Dates: First submitted 2021-01-20; First posted 2021-02-02 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Healthy Infants
MeSH Terms: interventions — Congresses as Topic

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- a2 Group (Active Comparator): The infant group consuming a2 Platinum® stage 1 infant formula
  Interventions: Other: a2 Platinum® stage 1 infant formula
- Control Group (Active Comparator): The infant group consuming conventional, A1 and A2 β-casein containing stage 1 infant formula
  Interventions: Other: Conventional, A1 and A2 β-casein containing stage 1 infant formula
- breast feeding (No Intervention)

INTERVENTIONS:
Other: a2 Platinum® stage 1 infant formula — Upon randomization (if not included in the breastfed group), each participant will be provided with up to 105 days' supply of the standardized formula and up to 28 days' supply of the allocated formula. Participants and study investigators will conduct the trial via a pre-determined randomization schedule.
  Arms: a2 Group
Other: Conventional, A1 and A2 β-casein containing stage 1 infant formula — Upon randomization (if not included in the breastfed group), each participant will be provided with up to 105 days' supply of the standardized formula and up to 28 days' supply of the allocated formula. Participants and study investigators will conduct the trial via a pre-determined randomization schedule.
  Arms: Control Group

SUMMARY:
This trial is a single-blind, randomized, controlled, parallel-designed trial to compare the effects of a2 Platinum® stage 1 infant formula versus conventional, A1 and A2 β-casein-containing stage 1 infant formula versus breastfeeding on crying, tolerance, gut health, and immune function.

DETAILED DESCRIPTION:
The protocol was updated from V8.2 to V9.1 and was approved by the Ethical Committee of Shanghai First Maternity and Infant Hospital, the main site. The major changes are: from "blind to participants" to "non-blind to participants"; from "Single-Centre" to "Multi-Centre"; number of subjects from "270" to "180"; trial period from "3 weeks" to "4 weeks"; and number of visits from "6" to "4".

ELIGIBILITY:
Inclusion Criteria:

1. 0-76 days of age after birth, inclusive (day of birth is considered day 0)
2. Singleton birth
3. Gestational age of 37-42 weeks (36 weeks and six days is considered 36 weeks gestational age)
4. Birth weight of 2,500 g to 4,500 g
5. Signed informed consent obtained for infant's participation in the survey
6. Parent or guardian of infant agrees not to enrol infant in another interventional clinical survey while participating in this survey
7. Parent or guardian agrees to formula-feed the baby as per the randomization schedule

For the formula-fed groups, participants in addition to the above-listed criteria, must also meet the following criterion:

- Parent or guardian agrees that the baby will be fed with standardized formula upon enrolment and switched to randomized formula at baseline (90-105 days of age)

For the breastfed group, participants in addition to the above-listed criteria, must also meet the following criterion:

- Parent or guardian agrees that the baby will be breast-fed

Exclusion Criteria:

1. Infant with inborn malformation and with hereditary and/or chronic and/or inborn diseases that could interfere with the survey (e.g. being unable to breast-feed or formula-fed)
2. Diseases jeopardizing intrauterine growth
3. Known or increased risk of IgE-mediated cow's milk protein allergy

   1. (i.e. one of the biological parents and/or siblings diagnosed with similar allergy,
   2. asthma, hay fever, etc.)
4. Infant with an acute infection or gastroenteritis at time of randomization
5. Evidence of feeding difficulties or formula intolerance, such as vomiting or poor intake at time of randomization
6. Participation in another clinical trial
7. Investigator's uncertainty about the willingness or ability of the parents to comply with the protocol requirements (including to fill in the diaries and to wait with introducing weaning foods until 4 months of age, and capability and willingness to do stool sample collection, handling, processing, and storage as instructed)
8. Infant is immunocompromised (according to a doctor's diagnosis of immunodeficiencies such as combined immunodeficiencies, DiGeorge Syndrome, Wiskott-Aldrich syndrome, severe congenital neutropenia and secondary immunodeficiencies linked to HIV infection, Down Syndrome or others) and children with known head/brain disease/injury such as microcephaly, macrocephaly or others

Exit Criteria:

1. Ineligibility (either arising during the trial or retrospectively having been overlooked at screening)
2. Significant protocol deviation
3. Significant non-compliance with product regimen or trial requirements
4. An adverse event (including one occurring before the start of the trial period) which requires discontinuation of the trial product or results in inability to continue to comply with trial procedures
5. Disease progression which requires discontinuation of the trial product or results in inability to continue to comply with trial procedures
6. Withdrawal of Consent
7. Lost to follow up
8. Weight at Visit 2 is <95% of birth weight [(weight at Visit 2÷birth weight) x 100 <95%]
9. Use of antibiotics, steroids or prebiotics/probiotics anytime between 14 days before baseline and trial completion
10. Participant whose mother has used any form of antibiotics or steroids while breastfeeding
11. More than 1 feed of formula milk per day for the breastfed group
12. More than 2 feeds of breast milk per day for the formula groups

Ages: 0 Days to 76 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-04-16 (Actual); Study Completion 2022-04-16 (Actual)

PRIMARY OUTCOMES:
Changes of crying frequency at each follow up visit compared to baseline | Visit 2 (baseline [90-105 days since birth]); Visit 3 (14 days after baseline); Visit 4 (28 days after baseline)
  Record frequency of crying (times/d)
Changes of crying duration at each follow up visit compared to baseline | Visit 2 (baseline [90-105 days since birth]); Visit 3 (14 day after baseline); Visit 4 (28 days after baseline)
  Record duration of crying (min)
Changes in fecal MPO levels at each follow up visit compared to baseline | Visit 2 (baseline [90-105 days since birth]); Visit 3 (14 day after baseline); Visit 4 (28 days after baseline)
  Record fecal MPO (in Unit) as markers of inflammation

SECONDARY OUTCOMES:
Changes in salivary cortisol levels at each follow up visit compared to baseline | Visit 2 (baseline [90-105 days since birth]); Visit 3 (14 day after baseline); Visit 4 (28 days after baseline)
  Record salivary cortisol (nmol/L) as markers of immune function
Changes in body length | Visit 2 (baseline [90-105 days since birth]); Visit 3 (14 days after baseline); Visit 4 (28 days after baseline)
  Differences in length gain (cm/d)
Changes in body weight | Visit 1 (screening/randomization); Visit 2 (baseline [90-105 days since birth]); Visit 3 (14 day after baseline); Visit 4 (28 days after baseline)
  Differences in weight gain (kg/d)
Changes in head circumference | Visit 1 (screening/randomization); Visit 2 (baseline [90-105 days since birth]); Visit 3 (14 day after baseline); Visit 4 (28 days after baseline)
  Differences in head circumference (cm/d)
Number of adverse events at each follow up visit compared to baseline | Visit 1 (screening/randomization); Visit 2 (baseline [90-105 days since birth]); Visit 3 (14 day after baseline); Visit 4 (28 days after baseline)
  Record number of adverse events as a measure of safety and tolerability
Abundance analysis of gut microflora species | Visit 2 (baseline [90-105 days since birth]); Visit 3 (14 days after baseline); Visit 4 (28 days after baseline)
  Differences in abundance of gut microflora species

CONTACTS AND LOCATIONS:
Overall Officials: Jiangqin Liu, MD, Principal Investigator — Shanghai First Maternity and Infant Hospital
Locations (5):
- China (5):
  - Nanjing Maternity and Child Health Care Hospital, Nanjing, Jiangsu
  - Second Hospital of Jilin University, Changchun, Jilin
  - Women & Children's Health Care Hospital of Linyi, China, Linyi, Shandong
  - Shanghai First Maternity and Infant Hospital, Shanghai, Shanghai Municipality
  - First Teaching Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No